CLINICAL TRIAL: NCT07057323
Title: Coronary Sinus Reducer For The Management Of Symptomatic Heart Failure With A Preserved Ejection Fraction Associated With Coronary Microvascular Dysfunction
Brief Title: Coronary Sinus Reducer For The Management Of Symptomatic Heart Failure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Amir Lerman, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-002292
Record Dates: First submitted 2025-06-26; First posted 2025-07-09 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Heart failure with a preserved ejection fraction (HFpEF) (Experimental): Subjects with diagnosed Heart failure with a preserved ejection fraction (HFpEF), non-obstructive Coronary Artery Disease (CAD), and have documented CMD.
  Interventions: Device: Coronary Sinus Reducer

INTERVENTIONS:
Device: Coronary Sinus Reducer — Subjects will have the Coronary Sinus Reducer implanted in their coronary sinus during a right heart catheterization procedure.

SUMMARY:
The purpose of this study is to evaluate the efficacy of CS Reducer implantation in patients with HFpEF and CMD on left ventricular filling pressures, specifically invasive measurement of PAWP during standardized exercise.

ELIGIBILITY:
Inclusion:

* Age ≥ 18
* Able to provide written informed consent and willing to participate in all required study follow-up assessments
* Clinical indicated coronary angiography with invasive CRT testing within 6 months prior to enrollment. Abnormal CFR of ≤ 2.5
* Symptomatic HFpEF defined by (PAWP>15mmHg at rest and /or PAWP>25 mmHg on exertion) during clinically performed Right heat catheterization with exercise performed within 6 months of enrollment or during screening visit (if not performed clinically in the last 6 months).
* Non-Obstructive CAD (≤ 50% stenosis in epicardial vessels and/or iFR>0.89 or FFR>0.8 in vessels with 50 to 70% stenosis)

Exclusion:

* History of left ventricular (LV) ejection fraction <50%
* Significant epicardial CAD (angiographic stenosis ≥70% or positive FFR or iFR in any major epicardial coronary artery
* Significant valvular heart disease (more than moderate regurgitation and or stenosis)
* Primary cardiomyopathies (hypertrophic, infiltrative or restrictive)
* Constrictive pericarditis
* Severe myocardial bridging
* Stiff left atrial syndrome
* Pregnancy
* Recent (with 3 months) acute coronary syndrome
* Subjects in Cardiogenic shock (systolic pressure<80mm/Hg)
* NYHA Class III or IV heart failure decompensated HF
* Mean right atrial pressure at rest >15 mmHg
* Anomalous or abnormal CS anatomy (e.g. tortuosity aberrant branch persistent left superior vena cava as demonstrated on angiogram
* CS diameter at the site of planned implantation greater than 13mm or less than 9.5 mm as measured by angiogram.
* Known severe reaction to required procedural medications
* Known allergy to stainless steel or nickel
* Magnetic Resonance Imaging (MRI) within 8 weeks after Reducer implantation
* Chronic renal failure (serum creatinine>2mg/dL)
* Severe chronic obstructive pulmonary disease (COPD) as indicated by forced expiratory volume in one second that is less than 55% of the predicted value or need for home daytime oxygen
* Pacemaker electrode/lead in the coronary sinus
* Moribund or with comorbidities limiting life expectancy to less than one year
* Current or past participation within a specified timeframe in another clinical trial, as warranted by the administration of this intervention.
* Inability or unwillingness of individual to give written informed consent.
* Additional factors deemed unsuitable for trial enrollment per discretion of the Principal Investigator
* Inmates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary Arterial Wedge Pressure (PAWP) at exercise | Baseline, 6 months
  Pulmonary Arterial Wedge Pressure (mmHg) is a measure of cardiac filling pressure. PAWP will be determined by a right heart catheterization at 20W exercise.

SECONDARY OUTCOMES:
Change in Kansas City Cardiomyopathy (KCCQ-12) | Baseline, 30 Days, 60 Days, 90 Days, 6 months
  KCCQ is a 12-item questionnaires that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. Scores were generated for each domain and scaled from 0 to 70, with 0 (worst) and 70 (the best possible status), where the higher score reflected better health status.
Change in Seattle Angina Questionnaire (SAQ) | Baseline, 30 Days, 60 Days, 90 Days, 6 months
  Seattle Angina Questionnaire (SAQ) is a 19-item questionnaire that assesses 5 different scales: physical limitation, anginal stability, anginal frequency, treatment satisfaction, and disease perception. A higher score indicates a worse health status.
Change in New York Heart Association (NYHA) classification | Baseline, 6 months
  New York Heart Association (NYHA) classification is used to classify patients into 4 categories based on their Heart Failure Symptoms. There are 4 classifications (1-4), a higher classification indicates a higher severity of Heart Failure symptoms.
Change in Canadian Cardiovascular Society (CCS) | Baseline, 30 Days, 60 Days, 90 Days, 6 months
  Canadian Cardiovascular Society (CCS) is a classification system (1-4) used to determine severity of angina pectoris. A higher classification indicates higher severity of angina pectoris.
Change in Borg maximal perceived exertion scores | Baseline, 6 months
  Borg CR10 Scale is a scale that ranges from 0-12. It is used to determine maximal perceived exertion. This will be measured at exercise during a right heart catheterization.
Change in maximum exercise capacity (VO2 max) during supine exercise testing | Baseline, 6 months
  Maximum exercise capacity (VO2 max) is the maximum oxygen absorbed during exercise. VO2 max will be determined at exercise during right heart catheterization and measured in ml/kg/min.
Change in transcardiac lactate release | Baseline, 6 months
  Transcardiac lactate release will be determined by blood sample and measured in mmol/L.
Change in transcardiac lactate uptake | Baseline, 6 months
  Transcardiac lactate uptake will be determined by blood sample and measured in mmol/L.
Change in Pulmonary Arterial Wedge Pressure (PAWP) at rest | Baseline, 6 months
  Pulmonary Arterial Wedge Pressure (mmHg) is a measure of cardiac filling pressure. PAWP will be determined by a right heart catheterization at rest.
Change in Pulmonary Arterial Pressure at rest | Baseline, 6 months
  Pulmonary Arterial Pressure is the measure of pressure that the heart uses to pump blood from the heart to the lungs. Pulmonary Arterial Pressure will be determined by a right heart catheterization at rest and measured in mmHg.
Change in Pulmonary Arterial Pressure at exercise | Baseline, 6 months
  Pulmonary Arterial Pressure is the measure of pressure that the heart uses to pump blood from the heart to the lungs. Pulmonary Arterial Pressure will be determined by a right heart catheterization at exercise and measured in mmHg.
Cardiac output | Baseline, 6 months
  Cardiac output (L/min) is the total volume of blood moved by the heart per minute. Cardiac output is measured during right heart catheterization at exercise using the Fick method.
Change in Right Atrial Pressure | Baseline, 6 months
  Right Atrial Pressure is the blood pressure in the right atrium.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No